CLINICAL TRIAL: NCT04615507
Title: Evaluation of a Daily Disposable Novel Multifocal Contact Lens in a Myopic Population
Brief Title: Evaluation of a Daily Disposable Novel Multifocal Contact Lens in a Myopic Population; Part 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CR-6413
Record Dates: First submitted 2020-10-29; First posted 2020-11-04 (Actual); Results first posted 2022-04-01 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Visual Acuity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Test/Control/Control (Experimental): Eligible subjects that are habitual soft contact lens wearers will be randomized to lens wear sequence, (Test/Control/Control)
  Interventions: Device: JJVC Investigational Multifocal Contact Lens; Device: Dailies Total 1® Multifocal Contact Lens
- Control/Test/Test (Experimental): Eligible subjects that are habitual soft contact lens wearers will be randomized to lens wear sequence, (Control/Test/Test)
  Interventions: Device: JJVC Investigational Multifocal Contact Lens; Device: Dailies Total 1® Multifocal Contact Lens

INTERVENTIONS:
Device: JJVC Investigational Multifocal Contact Lens — TEST Lens
Device: Dailies Total 1® Multifocal Contact Lens — CONTROL Lens

SUMMARY:
This is a 6-visit, subject-masked, multi-site, 2×3 crossover dispensing trial that will last approximately 2 - 4 months.

ELIGIBILITY:
Inclusion Criteria:

* Potential subjects must satisfy all the following criteria to be enrolled in the study:

  1. The subject must read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.
  2. The subject must appear able and willing to adhere to the instructions set forth in this clinical protocol.
  3. The subject must be at least 40 years of age and not greater than 70 years of age at the time of consent.
  4. Subjects must own a wearable pair of spectacles if required for their distance vision.
  5. The subject must be an adapted soft contact lens wearer in both eyes (i.e. worn lenses a minimum of 2 days per week for at least 6 hours per wear day, for 1 month or more duration).
  6. The subject must either already be wearing a presbyopic contact lens correction (e.g., reading spectacles over contact lenses, multifocal or monovision contact lenses, etc.) or, if not respond positively to at least one symptom on the "Presbyopic Symptoms Questionnaire" (Appendix E).
  7. The subject's distance spherical equivalent refraction must be in the range of -1.25 D to -3.75 D in each eye.
  8. The subject's refractive cylinder must be ≤0.75 D in each eye.
  9. The subject's ADD power must be in the range of +0.75 D to +2.50 D.
  10. The subject must have distance best corrected visual acuity of 20/20-3 or better in each eye.

      Exclusion Criteria:
* Potential subjects who meet any of the following criteria will be excluded from participating in the study:

  1. Currently pregnant or lactating.
  2. Any active or ongoing ocular or systemic allergies that may interfere with contact lens wear.
  3. Any active or ongoing systemic disease, autoimmune disease, or use of medication, which may interfere with contact lens wear. This may include, but not be limited to, diabetes, hyperthyroidism, Sjögren's syndrome, xerophthalmia, acne rosacea, Stevens-Johnson syndrome, and immunosuppressive diseases or any infectious diseases (e.g. hepatitis, tuberculosis).
  4. Any previous, or planned, ocular or intraocular surgery (e.g. radial keratotomy, PRK, LASIK, lid procedures, cataract surgery, retinal surgery, etc.).
  5. A history of amblyopia, strabismus or binocular vision abnormality.
  6. Use of any of the following medications within 2 weeks prior to enrollment: oral retinoids, oral tetracyclines, anticholinergics, systemic/topical steroids, oral phenothiazines. See section 9.1 for additional details regarding excluded systemic medications.
  7. Use of any ocular medication, with the exception of rewetting drops.
  8. History of herpetic keratitis.
  9. History of irregular cornea.
  10. History of pathological dry eye.
  11. Participation in any contact lens or lens care product clinical trial within 30 days prior to study enrollment.
  12. Employee or immediate family member of an employee of clinical site (e.g., Investigator, Coordinator, Technician).
  13. Any known hypersensitivity or allergic reaction to non-preserved rewetting drop solutions or sodium fluorescein.

      Exclusion Criteria after Baseline:
  14. Clinically significant (Grade 2 or greater) corneal edema, corneal vascularization, corneal staining, tarsal abnormalities or bulbar injection, or any other corneal or ocular abnormalities which would contraindicate contact lens wear.
  15. Entropion, ectropion, extrusions, chalazia, recurrent styes, glaucoma, history of recurrent corneal erosions.
  16. Any current ocular infection or inflammation.
  17. Any current ocular abnormality that may interfere with contact lens wear

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2020-10-09 (Actual); Primary Completion 2020-12-09 (Actual); Study Completion 2020-12-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Vue Optical Boutique, Jacksonville, Florida
  - Visual Eyes, Inc., Roswell, Georgia
  - Advanced Eye Care, Raytown, Missouri
  - Susquehanna Eye Care, Vestal, New York
  - ProCare Vision Centers, Granville, Ohio
  - West Bay Eye Associates, Warwick, Rhode Island

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu
URL: http://yoda.yale.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 71 subject were enrolled into this study. Of those enrolled, 68 were dispensed at least one study lens while 3 subjects failed to meet all eligibility criteria. Of those dispensed, 60 completed the study while 8 subjects were discontinued.
Groups:
- Test/Control/Control: Subjects that wore the Test lens in a bilateral fashion during period 1 and the Control lens during both the second and third study periods.
- Control/Test/Test: Subjects that wore the Control lens in a bilateral fashion during period 1 and the Test lens during the second and third study periods.
Period: Period 1
Arm/Group | Test/Control/Control | Control/Test/Test
Started | 34 | 34
Completed | 32 | 33
Not Completed | 2 | 1
Not completed — Covid-19 exposure | 2 | 1
Period: Period 2
Arm/Group | Test/Control/Control | Control/Test/Test
Started | 32 | 33
Completed | 30 | 31
Not Completed | 2 | 2
Not completed — Covid-19 exposure | 0 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Adverse Event | 0 | 1
Period: Period 3
Arm/Group | Test/Control/Control | Control/Test/Test
Started | 30 | 31
Completed | 30 | 30
Not Completed | 0 | 1
Not completed — Covid-19 exposure | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Test/Control/Control | Control/Test/Test | Total
Number analyzed (Participants) | 34 | 34 | 68
Age, Continuous [Mean (Standard Deviation); unit: Years]
  Age | 49.0 (4.72) | 52.0 (7.44) | 50.5 (6.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Sex: Female | 24 | 25 | 49
  Sex: Male | 10 | 9 | 19
Race/Ethnicity, Customized [Number; unit: participants]
  Black or African American | 1 | 3 | 4
  White | 33 | 31 | 64
Region of Enrollment [Number; unit: participants]
  United States | 34 | 34 | 68

OUTCOME MEASURES:

1. Primary Outcome: Visual Performance LogMAR
Description: Binocular visual performance on logMAR (Logarithm of Minimal Angle of Resolution) scale was evaluated at distance (4 meters), intermediate (64 centimeters) and near (40 centimeters) under high luminance high contrast lighting condition using ETDRS (Early Treatment Diabetic Retinopathy Study) charts. The room illuminance was required to be between 7.3 and 7.9 EV (394-597 lux). For Distance (4 meters), the acceptable range for the chart luminance was 10.5-10.7 EV (181 208 cd/m2). For Intermediate (64cm) and Near (40cm), the acceptable range for the chart luminance 10.8-11.1 EV (223-274 cd/m2). Letter-by letter results calculated the visual performance score for each chart read. logMAR scores closer to zero, or below zero, indicate a better visual acuity. A logMAR visual performance score of 0.0 is equivalent to Snellen visual acuity of 20/20.
Time Frame: 1-Week Follow-up within each wearing period
Population: All subjects that completed all study visits without a major protocol deviation impacting a primary endpoint.
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: Observations
Groups:
- Test: All subjects that wore the Test lens during any of the 3 study periods.
- Control: All subjects that wore the Control lens during any of the 3 study periods.
Arm/Group | Test | Control
Number analyzed (Participants) | 60 | 60
Number analyzed (Observations) | 90 | 90
logMAR
  Distance (4m) | -0.12 (0.108) | -0.13 (0.088)
  Intermediate (64cm) | -0.06 (0.089) | -0.04 (0.106)
  Near (40cm) | 0.08 (0.140) | 0.10 (0.136)
Statistical Analysis 1: Comparison: Test; Test type: Superiority — The superiority of the Test lens will be concluded if the upper confidence limit of the mean is below the predefined threshold +0.00 logMAR for Distance; Linear Mixed Model; Kenward and Roger Method was used for denominator degrees of freedom; Mean estimate = -0.132, 95% CI 2-sided [-0.180 to -0.083], Standard Error of Mean 0.0201
Statistical Analysis 2: Comparison: Test; Test type: Superiority — The superiority of the Test lens will be concluded if the upper confidence limit of the mean is below the predefined threshold +0.17 logMAR for Intermediate; Linear Mixed Model; Kenward and Roger Method was used for denominator degrees of freedom; Mean estimate = -0.066, 95% CI 2-sided [-0.115 to -0.017], Standard Error of Mean 0.0202
Statistical Analysis 3: Comparison: Test; Test type: Superiority — The superiority of the Test lens will be concluded if the upper confidence limit of the mean is below the predefined threshold +0.17 logMAR for Near; Linear Mixed Model; Kenward and Roger Method was used for denominator degrees of freedom; Mean estimate = 0.072, 95% CI 2-sided [0.022 to 0.121], Standard Error of Mean 0.0217

2. Secondary Outcome: Vision Scores
Description: Overall vision scores were assessed using the Contact Lens User Experience™ (CLUE) questionnaire. CLUE is a validated patient-reported outcomes (PRO) questionnaire to assess patient experience attributes of soft contact lenses (comfort, vision, handling, and packaging) in a contact-lens wearing population in the US, ages 18-65. Derived CLUE scores using Item Response Theory (IRT) follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response with a range of 0-120. The average CLUE vision score for each leans type was reported.
Time Frame: 1-Week Follow-up within each wearing period
Population: All subjects that completed all study visits without a major protocol deviation impacting a primary endpoint.
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Observations
Arm/Group | Test | Control
Number analyzed (Participants) | 60 | 60
Number analyzed (Observations) | 90 | 90
units on a scale | 59.72 (18.310) | 53.98 (15.108)
Statistical Analysis 1: Comparison: Test; Test type: Superiority — The superiority of the Test lens will be concluded if the lower confidence limit of the LSM is above the predefined threshold 32 points; Linear Mixed Model; Kenward and Roger Method was used for the denominator degrees of freedom; Least-square mean = 59.6, 95% CI 2-sided [52.3 to 66.8], Standard Error of Mean 3.05
Statistical Analysis 2: Comparison: Test vs Control; Test type: Non-Inferiority — The non-Inferiority of the Test lens relative to the Control will be concluded if the lower confidence limit of LSM difference is above -5 points; Linear Mixed Model; Kenward and Roger Method was used for the denominator degrees of freedom; Least-square mean difference = 5.5, 95% CI 2-sided [0.9 to 10.2], Standard Error of Mean 2.36 — LSM difference was calculated as Test minus Control

ADVERSE EVENTS:
Time Frame: Throughout the duration of the study; approximately 3 weeks per subject.
Arm/Group | Test | Control
All-Cause Mortality (participants affected / at risk) | 0/67 | 0/66
Serious Adverse Events (participants affected / at risk) | 0/67 | 0/66
Other Adverse Events (participants affected / at risk) | 0/67 | 0/66

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-05): https://cdn.clinicaltrials.gov/large-docs/07/NCT04615507/Prot_SAP_000.pdf